CLINICAL TRIAL: NCT02027701
Title: Multicenter, Open-label Extension Study to Investigate the Long-term Safety and Efficacy of IgPro20 in Maintenance Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) in Subjects Completing Study IgPro20_3003
Brief Title: Extension Study of Maintenance Treatment With Subcutaneous Immunoglobulin (IgPro20) for Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_3004; 2013-004157-24 (EudraCT Number)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP); Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IgPro20 (Experimental): 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for SC use administered SC weekly: 0.2 g/kg bw (low-dose IgPro20) for up to 48 weeks. Subjects who experience CIDP relapse on 0.2 g/kg IgPro20 will have an increase to 0.4 g/kg IgPro20 immediately and will continue on high-dose until they have completed a total of 48 weeks of IgPro20 treatment.
  Interventions: Biological: IgPro20

INTERVENTIONS:
Biological: IgPro20

SUMMARY:
This study is an extension study to the pivotal study IgPro20_3003 (NCT01545076). The purpose of this extension study is to investigate the long-term treatment of CIDP with IgPro20, with regard to safety and efficacy.

Subjects who have completed subcutaneous (SC) Week 25 or were successfully rescued from a CIDP relapse during the SC Treatment Period of pivotal study IgPro20_3003 (NCT01545076) will have the option to receive open-label low-dose IgPro20 (0.2 g/kg bodyweight [bw]) weekly for up to 48 weeks. Subjects relapsing on low-dose IgPro20 will either return to high-dose IgPro20 (0.4 g/kg) immediately or be discontinued, depending on investigator's judgment. Subjects returning to high-dose IgPro20 will continue on high-dose until they have completed a total of 48 weeks of IgPro20 treatment. If subjects do not successfully recover from CIDP relapse within 4 weeks, they will be withdrawn.

The treatment duration will be up to 48 weeks, followed by a completion visit (week 49).

ELIGIBILITY:
Inclusion Criteria:

* Subjects having completed the pivotal study IgPro20_3003 (SC Week 25) or successfully rescued from a CIDP relapse during the SC Treatment Period of pivotal study IgPro20_3003 (NCT01545076).
* Written informed consent for study participation obtained before undergoing any study-specific procedures.

Exclusion Criteria:

* Subject is unable to directly transition from study IgPro20_3003.
* New medical condition and/or social behavior (ie, alcohol, drug, or medication abuse) during participation in study IgPro20_3003 that in the judgment of the investigator could increase risk to the subject, interfere with the evaluation of investigational medicinal product, and/or conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ivo N. van Schaik, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (33):
- United States (5):
  - Site Reference 8400181, Birmingham, Alabama
  - Site Reference 8400167, Los Angeles, California
  - Site Reference 8400166, Kansas City, Kansas
  - Site Reference 8400169, New York, New York
  - Site Reference 8400182, Charlotte, North Carolina
- Australia (2):
  - Site Reference 0360017, Woolloongabba, Queensland
  - Site Reference 0360011, Fitzroy, Victoria
- Canada (2):
  - Site Reference 1240009, Toronto, Ontario
  - Site Reference 1240007, Greenfield Park, Quebec
- Czechia (2):
  - Site Reference 2030009, Hradec Králové
  - Site Reference 2030002, Hradec Králové
- Site Reference 2500022, Nice, France
- Germany (9):
  - Site Reference 2760052, Essen, North Rhine-Westphalia
  - Site Reference 2760069, Berlin
  - Site Reference 2760072, Berlin
  - Site Reference 2760049, Bochum
  - Site Reference 2760094, Essen
  - Site Reference 2760054, Hanover
  - Site Reference 2760055, Leipzig
  - Site Reference 2760047, Potsdam
  - Site Reference 2760039, Würzburg
- Site Reference 3800031, Milan, Italy
- Japan (6):
  - Site Reference 3920037, Tokorozawa, Saitama
  - Site Reference 3920035, Ube, Yamaguchi
  - Site Reference 3920038, Chiba
  - Site Reference 3920061, Kanagawa
  - Site Reference 3920040, Nagoya
  - Site Reference 3920065, Tokyo
- Site Reference 5280001, Amsterdam, Netherlands
- Spain (2):
  - Site Reference 7240011, Barcelona
  - Site Reference 7240010, Barcelona
- United Kingdom (2):
  - Site Reference 8260019, London
  - Site Reference 8260032, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- IgPro20: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin administered SC weekly at 0.2 g/kg, and subjects who experience CIDP relapse on 0.2 g/kg IgPro20 will have an increase to 0.4 g/kg IgPro20.
Period: Overall Study
Arm/Group | IgPro20
Started | 82
Completed | 66
Not Completed | 16
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 8
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- IgPro20: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for SC use administered SC weekly at 0.2 g/kg or 0.4 g/kg.
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.57 (13.224)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 70
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 7
  Netherlands | 1
  United States | 9
  Czechia | 2
  Japan | 10
  Italy | 8
  United Kingdom | 4
  Australia | 1
  France | 1
  Germany | 29
  Spain | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs) Per Infusion
Time Frame: Up to 49 weeks
Population: Safety Data Set (SDS): all subjects who received at least 1 dose of IgPro20 in this study.
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Groups:
- IgPro20: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for SC use administered SC weekly: 0.2 g/kg or 0.4 g/kg for up to 49 weeks.
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Number analyzed (Infusions) | 5553
Adverse events per infusion | 0.032

2. Secondary Outcome: Time to First CIDP Relapse
Description: Time to first CIDP relapse based on adjusted INCAT score, using the Kaplan-Meier estimator. Relapse is defined as an increase of at least 1 INCAT score point (except for the increase from 0 to 1 in the upper limb score only).
Time Frame: Up to 49 weeks
Population: Total Set: all subjects enrolled in the study, ie, the subject's informed consent was obtained. In the study protocol, this analysis set was referred to as the Intention-to-Treat Data Set.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Days | 266.0 [225.0 to NA] — The upper limit of the 95% confidence interval for the median time to relapse cannot be estimated, because the curve representing the upper confidence limit lies above 0.5.

3. Secondary Outcome: Change From Baseline in CIDP Total Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Score
Description: The INCAT score is a 10-point scale that covers the functionality of legs and arms, and has been successfully used to measure treatment effects in various CIDP studies. Scores for arm disability range from 0 ("No upper limb problems") to 5 ("Inability to use either arm for any purposeful movement"), and scores for leg disability range from 0 ("Walking not affected") to 5 ("Restricted to wheelchair, unable to stand and walk a few steps with help"). The INCAT (total) score is the sum of these 2 scores and ranges from 0 to 10. For the "adjusted" INCAT score, changes in the function of the upper limbs from 0 (normal) to 1 (minor symptoms) or from 1 to 0 were not recorded as deterioration or improvement because these changes are not considered clinically significant.
Time Frame: Baseline and up to 49 weeks
Population: Total Set
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20
Number analyzed (Participants) | 80
units on a scale | 0.0 [-3 to 6]

4. Secondary Outcome: Change From Baseline in Medical Research Council (MRC) Score
Description: An adapted version of the MRC sum score as published by Kleyweg and the RMC trial group was used. With the MRC sum score, the following 8 bilateral muscle pairs were assessed, and individual muscle scores as well as the sum score documented: Shoulder abduction; Elbow flexion; Wrist extension; Index finger abduction; Hip flexion; Knee extension; Foot dorsiflexion; Great toe dorsiflexion. The MRC sum score ranges from 0 (paralysis) to 80 (normal strength) points.
Time Frame: Baseline and up to 49 weeks
Population: Total Set
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20
Number analyzed (Participants) | 78
units on a scale | 0.0 [-23 to 18]

5. Secondary Outcome: Change From Baseline in Rasch-built Overall Disability Scale (R-ODS)
Description: The R-ODS is a recently published outcome measure that captures activity and social participation in subjects with Guillain-Barré Syndrome, CIDP, and monoclonal gammopathy of uncertain significance. The 24-item questionnaire covers a wide range of tasks of daily life that are each to be rated as "impossible to perform", "able to perform with difficulty", or "easy to perform" (scale of 0 - 2 points respectively). Items are sorted in order of increasing difficulty to perform, based on data from subjects with peripheral neuropathies (chronic inflammatory demyelinating polyneuropathy, Guillain-Barré Syndrome, or monoclonal gammopathy of uncertain significance) and subjects recruited at the university outpatient clinics of Rotterdam and Maastricht.
Time Frame: Baseline and up to 49 weeks
Population: Total Set
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20
Number analyzed (Participants) | 71
units on a scale | 0.0 [-76 to 33]

6. Secondary Outcome: Change From Baseline in Mean Grip Strength
Description: The hand-held Vigorimeter from Martin (Tuttlingen, Germany) is a device that measures the strength of small muscles in the hand, ie, grip strength. The subject squeezes a rubber bulb lying between the palm of the hand and the thumb and index fingers. The pressure is recorded via a rubber tube on a nanometer and expressed in kilopascal (kPa). At each assessment, the subject squeezes 3 times with each hand.
Time Frame: Baseline and up to 49 weeks
Population: Total Set
Measure: Median (Full Range); unit: kPa
Arm/Group | IgPro20
Number analyzed (Participants) | 79
kPa | -0.7 [-80 to 27]

7. Secondary Outcome: Percentage of Subjects With Adverse Events (AEs)
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro20
Number analyzed (Participants) | 82
percentage of subjects | 75.6

8. Secondary Outcome: Number of AEs by Severity Per Infusion
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Number analyzed (Infusions) | 5553
Adverse events per infusion
  Mild | 0.024
  Moderate | 0.006
  Severe | 0.002

9. Secondary Outcome: Percentage of Subjects With AEs by Severity
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: percentage of subjects
Groups:
- IgPro20: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for SC use administered SC weekly at 0.2 g/kg or 0.4 g/kg for up to 49 weeks.
Arm/Group | IgPro20
Number analyzed (Participants) | 82
percentage of subjects
  Mild | 62.2
  Moderate | 29.3
  Severe | 9.8

10. Secondary Outcome: Number of Causally Related AEs Per Infusion
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Number analyzed (Infusions) | 5553
Adverse events per infusion | 0.011

11. Secondary Outcome: Percentage of Subjects With Causally Related AEs
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro20
Number analyzed (Participants) | 82
percentage of subjects | 25.6

12. Secondary Outcome: Number of Serious AEs Per Infusion
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Groups:
- IgPro20: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for SC use administered SC weekly at 0.2 g/kg for up to 49 weeks.
Arm/Group | IgPro20
Number analyzed (Participants) | 82
Number analyzed (Infusions) | 5553
Adverse events per infusion | 0.001

13. Secondary Outcome: Percentage of Subjects With Serious AEs
Time Frame: Up to 49 weeks
Population: SDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro20
Number analyzed (Participants) | 82
percentage of subjects | 8.5

ADVERSE EVENTS:
Time Frame: Up to 49 weeks
Arm/Group | IgPro20
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 7/82
Other Adverse Events (participants affected / at risk) | 25/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=82)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 2 (2)
Nerve Compression (Nervous system disorders) | 1 (1)
Pulmonary Sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Immune system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Worsening of upper back pain secondary to fall. Non-treatment emergent SAE, occurring before first dose of IgPro20.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=82)
Infusion site swelling (Skin and subcutaneous tissue disorders) | 9 (11) — General disorders and administration site conditions
Infusion site erythema (Skin and subcutaneous tissue disorders) | 7 (9) — General disorders and administration site conditions
Infusion site swelling (Skin and subcutaneous tissue disorders) | 9 (11) — Local reactions
Infusion Site erythema (Skin and subcutaneous tissue disorders) | 7 (9) — Local reactions
Nasopharyngitis (Infections and infestations) | 11 (13)
Headache (Nervous system disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02027701/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02027701/SAP_001.pdf